CLINICAL TRIAL: NCT03371901
Title: Physical Therapy With Blood Flow Restriction Training to Enhance Recovery in Patients With Early Weight Bearing Restrictions After Knee Surgery: A Feasibility Study
Brief Title: Blood Flow Restriction Training in Patients With Weight Bearing Restrictions After Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Centre Nørrebro, City of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Linding Jakobsen, Research Physiotherapist, Health Centre Nørrebro, City of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHN
Record Dates: First submitted 2017-11-10; First posted 2017-12-13 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Cartilage, Articular; Tibial Meniscus Injuries
Keywords: Menisci, Tibial; Cartilage, Articular; Blood Flow Restriction Training; Resistance training; Physical Therapy Modalities; Feasibility Studies
MeSH Terms: conditions — Tibial Meniscus Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical therapy with BFR-LLST (Experimental)
  Interventions: Other: Physical therapy with BFR-LLST

INTERVENTIONS:
Other: Physical therapy with BFR-LLST — The criteria-based rehabilitation protocol for the patients with cartilage or meniscus repair may vary according to the surgical procedures.
  Patients will attend 5 individual treatments, and a 6-week supervised group-based rehabilitation program with BFR-LLST (Blood Flow Restriction - Low Load Strength Training) twice a week at the rehabilitation centre. Patient will be instructed to perform BFR-LLST 5 times a week in total (twice supervised, 3 times at home).
  During each BFR-LLST session, patients are encouraged to perform 4 sets of 30 repetitions, 15 repetitions, 15 repetitions, and 15 repetitions (or to fatigue in the final set), respectively.
  The exercise intervention will adhere to TIDieR (template for intervention description and replication).

SUMMARY:
After a cartilage or meniscus repair in the knee joint, the patients experience a pronounced and persistent decrease of knee-extension strength in the operated leg, which negatively affect patients' functional performance and quality of life. A possible novel exercise modality to increase muscle strength early is a moderate blood flow restriction with low-load strength training (BFR-LLST) exercise. BFR-LLST involves application of a wrapping device to restrict the blood flow to the muscle(s) during exercise. BFR- LLST requires much less load than traditional strength training and has shown to produce positive training adaptations such as muscle hypertrophy and strength in the lower extremity in healthy subjects and patients with a knee surgery. To our knowledge, early rehabilitation with BFR-LLST has never been investigated in a population with weight bearing restrictions, such as patients recovering from cartilage or meniscus repair in the knee joint. Fear of symptom exacerbation and adverse events have precluded BFR-LLST early after knee surgery. The purpose of this study is to examine the feasibility of 9 weeks of supervised rehabilitation with BFR-LLST early after cartilage or meniscus repair in the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a cartilage and/or meniscus repair in 1 or 2 knee(s).
* Patient is between 18 and 70 years.
* Patient is able to speak and understand Danish.
* Patient has given informed consent to participate in the study.

Exclusion Criteria:

* Patient has problems that severely limits ambulatory function from unstable orthopaedic (besides cartilage repair and meniscal fixation in the knee joint), neurological, vascular or cardiac conditions.
* Patient has a history of diagnosed major psychiatric disorder.
* Patient has a history of illicit drug use; be currently abusing alcohol or currently withdrawing from alcohol abuse.
* Patient has a history of endothelial dysfunction, peripheral vascular disease, hypertension, diabetes.
* Patient has a history of heart disease and deep vein thrombosis.
* Patient is pregnant.
* Patient has cancer (current diagnosis).
* Patient has an active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Thigh muscle hypertrophy assessed by thigh circumference, cm. | Change from baseline to the end of the 6-week rehabilitation program. Further assessments: Once a week during the 6-week rehabilitation program; 1 and 3 week(s) post-baseline, and 16 and 26 postoperative.
  Thigh circumference is assessed 15 cm. proximal from the basis of the patellae with a tape measure. The thigh circumference will be recorded to the nearest 0.1 cm, and assessed on both the operated and the non-operated leg.
  Being an exploratory feasibility study, the study is designed with a flat outcome structure with multiple evenly valued outcome measures. Thus, no primary and secondary outcome measure hierarchy exists, even though thigh muscle hypertrophy, assessed by thigh circumference, is presented as the primary outcome measure.

SECONDARY OUTCOMES:
Perceived exertion during exercise assessed by the Borg RPE scale (6-20)), points | Change from baseline to the end of the 6-week rehabilitation program. Further assessments: Once a week during the 6-week rehabilitation program; 1 and 3 week(s) post-baseline.
  The perceived exertion during BFR-LLST (Blood Flow Restriction - Low Load Strength Training) exercise is measured by using the Borg scale ranging from 6 (no exertion at all) to 20 (maximal exertion). The patients will be asked immediately after each set of BFR-LLST.
Adherence to the BFR-LLST (Blood Flow Restriction - Low Load Strength Training) protocol assessed by patient-reporting and assessor registration, numbers. | Change from baseline to the end of the 6-week rehabilitation program. Further assessments: Once a week during the 6-week rehabilitation program; 1 and 3 week(s) post-baseline.
  Adherence will be assessed during patient-reporting and assessor registration during visits at the rehabilitation centre. The number of training sessions, number of sets and repetitions, and training load will be registered.
Knee joint and quadriceps pain assessed by using 0-100-mm visual analog scale. | Change from baseline to the end of the 6-week rehabilitation program. Further assessments: Once a week during the 6-week rehabilitation program; 1 and 3 week(s) post-baseline.
  Assessment of pain is performed before (at rest), during and after (at rest) the BFR-LLST (Blood Flow Restriction - Low Load Strength Training) at the rehabilitation centre. Additionally, maximum knee joint and quadriceps pain during the rehabilitation program are assessed. The knee and quadriceps pain are assessed using a 0-100-mm visual analog scale with end points of "no pain" and "worst pain imaginable."
Knee joint swelling assessed by knee joint circumference, cm. | Change from baseline to 16 weeks postoperative. Further assessment: 26 weeks postoperative.
  Knee joint swelling of the operated leg is assessed by measuring the knee joint circumference 1 cm. proximal from the basis of the patellae with a tape measure.The knee joint circumference will be recorded to the nearest 0.1 cm.
Knee joint range of motion (ROM) assessed by goniometer, degrees | Change from baseline to 16 weeks postoperative. Further assessment: 26 weeks postoperative.
  Knee joint ROM of the operated leg is assessed using a large universal goniometer with the moveable arms pointing towards the greater trochanter and the lateral malleolus, respectively. Both the passive and active ROM are recorded to the nearest 1 degree.
Maximum isometric knee extension and flexion muscle strength at 60 degrees knee flexion assessed by a hand-held dynamometer in Nm/kg, (Newton*meter)/kg body weight | 26 weeks postoperative.
  The isometric muscle strength will be assessed using a hand-held dynamometer (MicroFET2 Hoggan Health Technologies Inc, UT, USA) on both the operated and non-operated leg.
Self-reported function and knee-related quality of life are assessed by using the Knee Injury and Osteoarthritis Outcome Score (KOOS), points | Change from baseline to 16 weeks postoperative. Further assessment: 26 weeks postoperative.
  The Knee injury and Osteoarthritis Outcome Score (KOOS) includes subscales of symptoms, pain, activities of daily living, function in sport/recreation, and knee-related quality of life. A score in points for each subscale will be calculated, and it ranges from 0 (worst score) to 100 (best score).
Self-reported patient-specific functional change is assessed by the Patient-Specific Functional Scale (PSFS) in points | Change from baseline to 16 weeks postoperative. Further assessment: 26 weeks postoperative.
  Patients are asked to identify 3 to 5 activities; they are having difficulty with as a result of their current problem. Each activity is scored on a 0 (unable to perform activity) to 10 (able to perform activity at same level as before injury or problem) points numeric rating scale. An average Patient-Specific Functional Scale (PSFS) score is calculated and can vary from 0 to 10, with higher scores representing higher levels of lower extremity functional status.

OTHER OUTCOMES:
Adverse events are assessed by patient-reporting and assessor registration. | Each visit from baseline to 26 weeks postoperative.
  All adverse events occurring while the patient is enrolled in the study will be documented regardless of its relation to the exercise intervention, operation or occurrences not related to the study. The number of possible adverse events are summed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Linding Jakobsen Jakobsen, PhD, Principal Investigator — Section for Orthopaedic & Sports Rehabilitation (SOS-R) Health Centre Nørrebro, City of Copenhagen, Denmark
Locations (1):
- Section for Orthopaedic & Sports Rehabilitation (SOS-R), Health Centre Nørrebro, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jakobsen TL, Thorborg K, Fisker J, Kallemose T, Bandholm T. Blood flow restriction added to usual care exercise in patients with early weight bearing restrictions after cartilage or meniscus repair in the knee joint: a feasibility study. J Exp Orthop. 2022 Oct 4;9(1):101. doi: 10.1186/s40634-022-00533-4. PMID 36192606